CLINICAL TRIAL: NCT03597594
Title: Haplocompatible Transplant Using TCRα/β Depletion Followed by CD45RA-Depleted Donor Lymphocyte Infusions for Severe Combined Immunodeficiency (SCID)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCIDBMT
Record Dates: First submitted 2018-06-19; First posted 2018-07-24 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Severe Combined Immunodeficiency
Keywords: Severe Combined Immunodeficiency; SCID; TCRα/β/CD19-depleted graft; CD45RA-depleted DLI; Graft-Versus-Host-Disease; Transplant
MeSH Terms: conditions — Severe Combined Immunodeficiency; Graft vs Host Disease | interventions — Antilymphocyte Serum; thymoglobulin; Busulfan; fludarabine; fludarabine phosphate; Thiotepa

STUDY DESIGN:
Intervention Model Description: Patients with SCID will receive TCRα/β-CD19 -depleted graft followed by CD45RA-depleted DLI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- TCRα/β/CD19-depleted SCT (Active Comparator): A preparative regimen based on the type of SCID will be given followed by infusion of donor cells. Cells for infusion are prepared using the CliniMACS System
  Regimen 1 - IL2RG, JAK 3 (Haplocompatible) and all MSD
  ATG (rabbit) IV Days -9 -8 and -7, Rest Days -6 and -5, Busulfan IV Days -4, -3, and -2, Rest Day -1, TCRα/β/CD19-depleted SCT, Day 0
  Regimen 2 - RAG1, RAG2 (Haplocompatible)
  ATG (rabbit) IV Days -9 -8 and -7, Fludarabine IV Days -7, -6, -5 and -4, Busulfan IV Days -5, -4 and -3, Thiotepa IV twice daily, Day -2, Rest Day -1, TCRα/β/CD19-depleted SCT, Day 0
  Regimen 3 - ADA, IL7R, CD45 deficiency, CD3 subunits (Haplocompatible)
  ATG (rabbit) IV Days -9 -8 and -7, Fludarabine IV Days -7, -6, -5 and -4, Busulfan: IV Days -4, -3 and -2, Rest Day -1, TCRα/β/CD19-depleted SCT, Day 0
  Interventions: Drug: Anti-thymocyte globulin (rabbit); Drug: Busulfan; Drug: Fludarabine; Drug: Thiotepa; Device: CliniMACS
- Donor Lymphocyte Infusions (Experimental): Phase I:
  On the Phase I portion of the study, up to 4 different dose levels will be evaluated: Dose level -1, Dose ≥0.1 to ≤0.3; Dose level 1, Dose >0.3 to ≤0.56; Dose level 2, Dose >0.56 to ≤1.8; Dose level 3, Dose >1.80 to ≤3.0
  Dosing is determined based on the number of CD3+CD45RA-cells/kg and the patient weight in kilograms.
  Phase II:
  Participants will receive the Phase I determined maximum tolerated dose (MTD) of DLI.
  Cells for infusion are prepared using the CliniMACS System.
  Interventions: Device: CliniMACS; Other: Donor Lymphocyte Infusion

INTERVENTIONS:
Drug: Anti-thymocyte globulin (rabbit) — given intravenously
  Other Names: Thymoglobulin®; rabbit ATG
  Arms: TCRα/β/CD19-depleted SCT
Drug: Busulfan — given intravenously
  Other Names: Myleran; Busulfex
  Arms: TCRα/β/CD19-depleted SCT
Drug: Fludarabine — given intravenously
  Other Names: Fludara
  Arms: TCRα/β/CD19-depleted SCT
Drug: Thiotepa — given intravenous infusion
  Other Names: TESPA; TSPA
  Arms: TCRα/β/CD19-depleted SCT
Device: CliniMACS — The mechanism of action of the CliniMACS Cell Selection System is based on magnetic-activated cell sorting (MACS). The CliniMACS device is a powerful tool for the isolation of many cell types from heterogeneous cell mixtures, (e.g. apheresis products). These can then be separated in a magnetic field using an immunomagnetic label specific for the cell type of interest, such as CD3+ human T cells.
  Other Names: Cell Selection System
Other: Donor Lymphocyte Infusion — given intravenous infusion
  Other Names: DLI
  Arms: Donor Lymphocyte Infusions

SUMMARY:
Infants with severe combined immunodeficiency (SCID) have a profound decrease in number and function of immune cells, and therefore remain highly vulnerable to infection. If not corrected this often leads to death. Hematopoietic cell transplantation (HCT) from matched sibling donor is the standard treatment for these patients, unfortunately though; most SCID patients lack a sibling donor. Building upon experience and existing data, the investigators are proposing a trial the goals of which are: to provide a conditioning regimen that is well tolerated, and provision of immune cells that altogether should establish rapid immune recovery providing protection from life threatening infections without increasing the risk of dangerous Graft-Versus-Host-Disease.

Primary Objectives

1. To evaluate the safety of a TCRα/β/CD19-depleted graft with CD45RA-depleted DLI in infants with SCID
2. To estimate overall survival at 1 year post transplantation

Exploratory Objectives

1. To evaluate the significant donor T cell reconstitution of a TCRα/β/CD19 depleted graft with CD45RA-depleted DLI at 1 year (+/-2 weeks).
2. To evaluate engraftment at day 30, 100, month 6, and years 1 to 10 post HCT.
3. To evaluate B cell reconstitution at years 1 to 10 post HCT.
4. To evaluate biomarkers of immune reconstitution at day 30, 60 100, month 6 and years 1 to 10; e.g. immunophenotype (including epigenetic profiling) of T, B, and NK cells, and assays to determine their function.
5. To evaluate clinical outcomes, post HCT.
6. To define the incidence and severity of acute (at day 100, month 6), and chronic (month 6, 12, 24) GVHD following HCT.

DETAILED DESCRIPTION:
In this study, the investigators propose to investigate T and B cell recovery using peripheral blood manipulation that removes potentially Graft-Versus-Host-Disease (GVHD) inducing α/β and CD45RA+ T cells, while still providing potentially beneficial donor γδ and memory T cells.

Donors will undergo a standard hematopoietic progenitor cell (HPC) mobilization regimen consisting of 5 days of G-CSF given subcutaneously at 10 micrograms/kilogram. The graft will be collected by leukapheresis on days 5 and if needed 6 of G-CSF. The HPC product(s) will be T-cell depleted (TCD) using the investigational CliniMACS device.

The initial HPC product(s) will be split into two portions; one portion will be used for TCR TCRαβ/CD19 depletion and the second portion for CD45depleted DLI product.

1. TCRα/β/CD19-depleted stem cell transplant: All participants will undergo a preparative regimen based on the type of Severe Combined Immunodeficiency (SCID) they have. This is followed by infusion of TCRα/β/CD19-depleted donor cells (with the exception of participants who undergo matched sibling donor HCT).
2. Donor Lymphocyte Infusion (CD45depleted DLI product): Participants, other than those who undergo matched sibling HCT transplant, will receive one dose of CD45RA depleted DLI infusion post TCRα/β/CD19-depleted graft infusion.

During the Phase I portion of the study, up to 4 different dose levels of CD45depleted DLI product will be evaluated.

On the Phase II portion of the study, all participants will receive the Phase I determined maximum tolerated dose (MTD) of DLI.

Participants on both the Phase I and Phase II portions of the study that are unable to receive protocol defined dosing of DLI due to insufficient dose generated will be eligible to receive the entirety of the generated product.

ELIGIBILITY:
Inclusion Criteria - Transplant Recipient

* Age ≥2 months old at the time of chemotherapy administration
* A proven mutation as defined by direct sequencing of patient DNA
* Has a suitable matched sibling donor or matched unrelated donor (8/8) or single haplotype matched (≥3 of 6) family member donor
* Patient must fulfill pre-transplant evaluation:
* Left ventricular ejection fraction >40% and no evidence of uncorrected congenital malformation with clinical symptomatology
* Creatinine clearance (CrCl) or glomerular filtration rate (GFR) ≥ 50 ml/min/1.73m2 or serum Creatinine ≤1.2mg/dL
* Resting pulse oximetry ≥90% on room or ≥95% on oxygen supplementation
* Lansky (age-dependent) performance score ≥50
* Bilirubin ≤3 times the upper limit of normal for age
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 5 times the upper limit of normal for age

Exclusion Criteria - Transplant Recipient

* Positive for HIV infection by genome PCR
* Presence of active malignancy
* A social situation indicating that the family may not be able to comply with protocol procedures and recommended medical care
* Presence of a medical condition indicating that survival will be dismal such as the requirement for mechanical ventilation, severe failure of a major organ system, or evidence of a serious, progressive infection that is refractory to medical therapy

Inclusion Criteria - Matched Sibling Donor and Haplocompatible Donor

* Fully matched sibling donor (8/8), or matched unrelated donor (8/8), or at least single haplotype matched (≥3 of 6) family member
* At least 1 year old (MSD) and at least 18 years of age (Haplocompatible)
* HIV negative
* Not pregnant as confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment (if female)
* Not breast feeding
* Regarding donation eligibility, is identified as either:

  * Completed the process of donor eligibility determination as outlined in 21 CFR 1271 and agency guidance; OR
  * Does not meet 21 CFR 1271 eligibility requirements, but has a declaration of urgent medical need completed by the principal investigator or physician sub-investigator per 21 CFR 1271

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of treatment related deaths | 42 days post DLI
  Treatment related deaths will be considered as one of the primary measures to evaluate the safety of a TCRα/β/CD19-depleted graft with CD45RA-depleted DLI in infants with SCID. Number of patients with treatment related deaths will be provided.
Number of overall grade 3-4 acute Graft-Versus-Host-Disease (GVHD) | 42 days post DLI
  Overall grade 3-4 acute GVHD events will be considered as one of the primary measures to evaluate the safety of a TCRα/β/CD19-depleted graft with CD45RA-depleted DLI in infants with SCID. Acute 3-4 GVHD events will be evaluated using established staging/grading criteria and expert consensus guidelines. Number of patients with overall grade 3-4 acute GVHD will be provided.
Overall Survival(OS) | 1 year post transplant
  To estimate OS at 1 year post transplantation. OS is defined as time from transplantation to death due to any cause. Patients who are alive at the time of analysis will be censored. Based on sample size, either binomial proportion or Kaplan-Meier analysis will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Ewelina Mamcarz, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols